CLINICAL TRIAL: NCT07133321
Title: The Effectiveness of Multi-pronged Interventions to Improve Institutional Delivery in South Ethiopia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Yves Jacquemyn (Other)
Collaborators: Flemish Interuniversity Council (VLIR) (Network); Arba Minch University (Other)
Responsible Party: Sponsor-Investigator, Prof Yves Jacquemyn, Dr. Professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: AMU-IUC-P3
Record Dates: First submitted 2025-07-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Maternal Health; Gender
Keywords: Institutional delivery; postnatal care; Husband involvement; husband equitable gender norm; Respectful maternal care; helping mothers survive
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Intervention Model Description: This study is a cluster randomized controlled trial conducted in Southern Ethiopia. Clusters (communities) are randomly assigned to one of four parallel arms: (1) husband group education only, (2) health worker helping mother survive + RMC training only, (3) both husband education and health worker training combined, or (4) control group receiving standard care. The husband education focuses on increasing knowledge and involvement in birth preparedness, shared decision-making, and responsibility sharing. The health worker training enhances skills in managing childbirth emergencies and providing culturally sensitive and respectful care. Randomization is done at the cluster level to avoid contamination. The study is open-label without masking due to the nature of interventions. The primary aim is to evaluate the effect of these interventions on improving maternal health service utilization, including institutional delivery and postpartum care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Husband Group Education Only (Experimental): group sessions for husbands focused on birth preparedness, shared decision-making, and shared responsibility to support maternal health service utilization.
  Interventions: Behavioral: Husband Group Health education.
- helping mother survive + RMC Training Only (Experimental): training for health professionals to enhance skills in managing childbirth emergencies, making referrals, and providing culturally sensitive, woman-centered care.
  Interventions: Behavioral: Helping Mothers Survive + RMC
- Combined Intervention (Experimental): both husband education and helping mother survive + RMC Training implemented concurrently.
  Interventions: Behavioral: Husband Group Health education.; Behavioral: Helping Mothers Survive + RMC
- Control Group (No Intervention): no additional interventions beyond standard care.

INTERVENTIONS:
Behavioral: Husband Group Health education. — The community-based husband group health education will target expectant fathers with pregnant partners. It will focus on reshaping gender-related attitudes and beliefs, promoting caregiving best practices, preventing violence against women, and improving men's involvement in maternal health. The intervention will comprise group sessions with 20 participants each, conducted over three sessions lasting 2.5 hours each, with a 15-day interval between sessions. The sessions will cover key topics, including recognizing obstetric danger signs, preparing for childbirth, fostering men's engagement in maternal health, advocating nonviolence and shared responsibility, and encouraging joint decision-making.
  Arms: Combined Intervention; Husband Group Education Only
Behavioral: Helping Mothers Survive + RMC — The "Helping Mothers Survive" training is designed by Jhpiego, an affiliate of Johns Hopkins University, in collaboration with global health partners, including the World Health Organization (WHO), Laerdal Global Health, and the International Confederation of Midwives (ICM) for healthcare professionals involved in childbirth care focusing on saving lives at birth in low-resource settings. This on-site training will use realistic simulations to enhance skills in identifying and managing key causes of maternal mortality, such as postpartum hemorrhage and preeclampsia, starting with essential labor care. The program employs the MamaNatalie birthing simulator, a low-tech realistic tool for hands-on practice developed by Laerdal Global Health. MamaNatalie features a model uterus with a neonate, placenta, and umbilical cord, enabling simulations of postpartum hemorrhage, breech delivery, vacuum-assisted birth, and normal labor.
  Arms: Combined Intervention; helping mother survive + RMC Training Only

SUMMARY:
This study aims to improve the health and safety of mothers during pregnancy and childbirth by working closely with their husbands. In many communities in Ethiopia, husbands play an important role in decisions about where women give birth.

The study involves educating husbands in group sessions to help them understand how to support their wives during pregnancy, prepare for childbirth, recognize danger signs, and encourage giving birth in health centers where skilled care is available.

At the same time, some health workers receive training to improve their ability to handle childbirth emergencies and provide respectful, culturally sensitive care.

Communities are divided into groups that receive either husband education, health worker training, both, or no additional support. The study will see which approach helps more women deliver safely in health centers and receive care after birth.

By involving husbands and improving health worker skills, this study hopes to support mothers better and improve outcomes for families.

DETAILED DESCRIPTION:
This study is conducted in Southern Ethiopia to improve the utilization of maternal health services, helping more women access safe childbirth and postnatal care. Many women face challenges in using health facilities for delivery, which can increase risks for mothers and babies. The study tests two key interventions that support mothers by involving both their families and health workers.

1. Husband Group Education:

   Since husbands often influence decisions about childbirth, this intervention provides group education sessions for husbands. These sessions focus on:

   Supporting their wives during pregnancy and childbirth.

   Preparing for birth and recognizing danger signs.

   Encouraging facility-based delivery where skilled care is available.

   Promoting shared decision-making and responsibility sharing between husbands and wives around pregnancy and childbirth.

   By increasing husbands' knowledge and encouraging joint responsibility, the study aims to improve the use of maternal health services by women.
2. Health Worker Training on Helping mother survive integrated RMC:

This intervention improves health workers' skills at local health facilities in Southern Ethiopia to:

Manage common childbirth emergencies.

Provide timely referrals and emergency care.

Deliver culturally sensitive and woman-centered care.

Enhance overall quality of care, making health facilities more effective and trusted.

The study uses a cluster randomized controlled trial design with four groups to compare the effects of these interventions:

Husband group education only,

Health worker training only,

Both husband education and health worker training,

No intervention (control group).

The primary goal is to identify which intervention best increases the number of women who give birth at health facilities and receive postnatal care. Secondary goals include improving husbands' knowledge and attitudes about birth preparedness, gender roles, and shared responsibilities, as well as enhancing health workers' knowledge and skills.

Overall, this study seeks to find effective ways to increase maternal health service utilization by fostering husband involvement and strengthening health system readiness, contributing to safer childbirth and healthier families in Southern Ethiopia

ELIGIBILITY:
Inclusion Criteria:

A husband whose wife is under 27 weeks of gestation

* A husband whose wife had a previous baby within 5 years
* A husband who lives with his wife together
* A husband who has lived with his wife in the selected cluster for at least six months

Exclusion Criteria:

-

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 1680 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
institutional delivery | 8 months/ 37 weeks
  Proportion of women who delivered in a health facility, institutional delivery refers to childbirth in a health facility, such as a hospital or health center, where skilled birth attendants are available to manage normal deliveries and handle complications that may occur
Maternal postnatal care | 8 months/37 weeks
  Proportion of mothers receiving at least one postnatal care visit within 6 weeks postpartum. The care given to the mother right after delivery and during the six weeks following childbirth (having at least one maternal postpartum care within six weeks of delivery)

SECONDARY OUTCOMES:
Husband's involvement in maternal health | 8 months/37 weeks
  Husband involvement was measured using the 21-item structured questionnaire adapted from the Global Framework for Assessing Male Participation in Maternal Health (Delphi method). Total scores range from 0 to 21. The mean score will be reported, and husbands will also be classified into three categories: low, moderate, and high involvement based on the sample distribution.
knowledge of obstetric danger signs and birth preparedness | 8 months/ 37 weeks
  Proportion that knew the danger signs of pregnancy, childbirth and postpartum period. Knowledge of obstetric danger signs includes identifying complications that may arise during pregnancy, labor and childbirth, and the postpartum period. Similarly, knowledge of birth preparedness involves knowing the planning for key aspects of safe delivery, such as arranging transportation, saving money, identifying blood donors, selecting a skilled provider, Identifying the place of delivery, Identifying someone to provide support, and preparing essential supplies like clean sheets, baby clothes, and sanitary items. Husbands who correctly listed at least three danger signs will be classified as having good awareness, while those who listed fewer than three will be classified as having poor awareness.
Gender-equitable attitude | 8 months/ 37 weeks
  Assesses attitudes toward gender norms, particularly in areas such as relationships, domestic responsibilities, reproductive health, and gender-based violence. For each participant, responses to the GEM scales were added together to form composite discrete variables that were categorized into high inequity = 24-39, Moderate inequity = 40-55, and low inequity = 56-72. Participants responded: Totally Agree =1; Partially Agree =2, or Do Not Agree=3 for each of the items of GEM scale Score.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Jacquemyn, Professor, Gynecology, Study Chair — Universiteit Antwerpen; Veerle Draulans, Professor, sociology, Study Chair — KU Leuven; Jean-pierre vangeertruyden, Professor, infectious disesase, Study Chair — Universiteit Antwerpen
Locations (1):
- Arba Minch university, Arba Minch, Southern Nations Nationalities Regional State, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided